CLINICAL TRIAL: NCT05829551
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics of RAY1216 and the Effect of Food on RAY1216 Pharmacokinetics in Healthy Adult Participants
Brief Title: The Safety, Tolerability and Pharmacokinetics Study of RAY1216 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAY1216-22-01
Record Dates: First submitted 2023-04-03; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 (Coronavirus Disease 2019)
MeSH Terms: conditions — COVID-19 | interventions — Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- RAY1216 dose 1 (Experimental): SAD
  Interventions: Drug: RAY1216 dose 1
- RAY1216 dose 2 (Experimental): SAD
  Interventions: Drug: RAY1216 dose 2
- RAY1216 dose 3 (Experimental): SAD
  Interventions: Drug: RAY1216 dose 3
- RAY1216 dose 4（DDI） (Experimental): drug-drug interaction
  Interventions: Drug: RAY1216 dose 4 &ritonavir
- RAY1216 dose 5 (Experimental): MAD
  Interventions: Drug: RAY1216 dose 5
- RAY1216 dose 6 (Experimental): MAD
  Interventions: Drug: RAY1216 dose 6
- RAY1216 dose 7 (Experimental): MAD
  Interventions: Drug: RAY1216 dose 7
- RAY1216 dose 8 (Experimental): MAD
  Interventions: Drug: RAY1216 dose 8
- RAY1216 dose 9（food effect） (Experimental): food effect on single dose
  Interventions: Drug: RAY1216 dose 9
- RAY1216 dose 10（food effect） (Experimental): food effect on single dose
  Interventions: Drug: RAY1216 dose 10

INTERVENTIONS:
Drug: RAY1216 dose 1 — RAY1216 dose 1 or Placebo
  Arms: RAY1216 dose 1
Drug: RAY1216 dose 2 — RAY1216 dose 2 or Placebo
  Arms: RAY1216 dose 2
Drug: RAY1216 dose 3 — RAY1216 dose 3 or Placebo
  Arms: RAY1216 dose 3
Drug: RAY1216 dose 4 &ritonavir — RAY1216 dose 4 &ritonavir or Placebo
  Arms: RAY1216 dose 4（DDI）
Drug: RAY1216 dose 5 — RAY1216 dose 5 or Placebo
  Arms: RAY1216 dose 5
Drug: RAY1216 dose 6 — RAY1216 dose 6 or Placebo
  Arms: RAY1216 dose 6
Drug: RAY1216 dose 7 — RAY1216 dose 7 or Placebo
  Arms: RAY1216 dose 7
Drug: RAY1216 dose 8 — RAY1216 dose 8 or Placebo
  Arms: RAY1216 dose 8
Drug: RAY1216 dose 9 — RAY1216 dose 9 or Placebo with high fat meal
  Arms: RAY1216 dose 9（food effect）
Drug: RAY1216 dose 10 — RAY1216 dose 10 or Placebo with high fat meal
  Arms: RAY1216 dose 10（food effect）

SUMMARY:
This is double-blind,randomized, single and multiple dose trial to evaluate the pharmacokinetics(PK), safety, tolerability and drug-drug interaction of RAY1216, and the effect of food on RAY1216 Pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of a dated Informed Consent Form (ICF) indicating that the subject has been informed of all the relevant aspects(including adverse events) of the trial prior to enrollment.
2. Subjects must be willing and able to adhere to the visit schedule and protocol requirements and be available to complete the study.
3. Subjects (including partners) must use reliable methods of contraception during the study and until 6 months following the last dose of investigational product.
4. Males and female subjects between 18-50 years (Both inclusive). Body weight is no less than 50 kg in males and no less than 45 kg in females. Body mass index (BMI) 18≤BMI≤28 kg/m2; BMI is determined by the following equation: BMI = weight/height2 (kg/m2).
5. Physical condition and vital signs: Normal or abnormality has no clinical significance.

Exclusion Criteria:

1. Known hypersensitivity and/or allergy to some drugs and food, especially for the composition that is similar to the investigative product;
2. The average daily smoking are more than 5 cigarettes within 3 months prior to screening.
3. Known history of drug or alcohol abuse.(defined as consumption of 14 units of alcohol per week: 1 unit = 285 ml of beer; or the equivalent of 25 ml of spirit, or 100 ml of wine )
4. Subjects who donated blood or bleeding profusely (> 400 mL) in the 3 months preceding study screening.
5. Dysphagia or any medical history in gastrointestinal that interferes with the absorption of drugs, include a history of frequent nausea or vomit causes by any etiology.
6. History or presence of any disease or condition known to increase the risk of bleeding , eg. acute gastritis, duodenal ulcer, etc.
7. Participated in another clinical research study and received any investigational products within 3 months prior to dosing.
8. History of having any special food (including dragon fruit, mango, grapefruit, etc.), strenuous exercises, or other factors may interfere with the absorption, distribution, metabolism, or excretion of drug within 7 days prior to screening.
9. Inability to consume the food provided in the study ( a high fat diet).This requirement only applies to subjects under fed condition.
10. Presence of clinically significant abnormalities in ECG or QTcF>450ms
11. Subjects who may not complete the study for other reasons or should not be included in the study in the opinion of the investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Number and severity of participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events(SAE) in single ascending dose | Day 1 to Day 5
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported
Number and severity of participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events(SAE) in multiple ascending dose | Day 1 to Day 9
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported
Number and severity of participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events(SAE) in DDI part | Day 1 to Day 15
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported
Number and severity of participants with Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events(SAE) in food effect part | Day 1 to Day 21
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported

SECONDARY OUTCOMES:
To determine the effect of food on the PK of RAY1216 single dose(Cmax) | Day 1 to Day 21
To investigate the effect of Ritonavir on the pharmacokinetics of RAY1216(Cmax) | Day 1 to Day 15
To determine the single and multiple oral dose pharmacokinetic profiles of RAY1216(Cmax) | Day 1 to Day 9
To determine the effect of food on the PK of RAY1216 single dose(AUC0-∞) | Day 1 to Day 21
To investigate the effect of Ritonavir on the pharmacokinetics of RAY1216(AUC0-∞) | Day 1 to Day 15
To determine the single and multiple oral dose pharmacokinetic profiles of RAY1216(Cmin) | Day 1 to Day 9

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Jilin, China

REFERENCES:
- [Derived] Hu Y, Li H, Wang K, Wu D, Zhang H, Ding Y, Wu J, Ye S, Peng Y, Liu L. Single- and multiple-dose pharmacokinetics and safety of the SARS-CoV-2 3CL protease inhibitor RAY1216: a phase 1 study in healthy participants. Antimicrob Agents Chemother. 2025 Mar 5;69(3):e0145024. doi: 10.1128/aac.01450-24. Epub 2025 Jan 31. PMID 39887246